CLINICAL TRIAL: NCT03568461
Title: A Phase II, Single Arm, Multicenter Open Label Trial to Determine the Efficacy and Safety of Tisagenlecleucel (CTL019) in Adult Patients With Refractory or Relapsed Follicular Lymphoma
Brief Title: Efficacy and Safety of Tisagenlecleucel in Adult Patients With Refractory or Relapsed Follicular Lymphoma
Acronym: ELARA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCTL019E2202; 2017-004385-94 (EudraCT Number); 2023-508127-13-00 (Registry Identifier: EU CTIS)
Record Dates: First submitted 2018-05-24; First posted 2018-06-26 (Actual); Results first posted 2022-07-22 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Follicular Lymphoma
Keywords: Refractory or relapsed Follicular Lymphoma; Refractory; Relapsed; Follicular lymphoma; CTL019; Tisagenlecleucel; Chimeric antigen receptor; CAR19; CAR-T
MeSH Terms: conditions — Lymphoma, Follicular; Recurrence | interventions — tisagenlecleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTL019 (Experimental): All patients who received tisagenlecleucel infusion.
  Interventions: Biological: tisagenlecleucel

INTERVENTIONS:
Biological: tisagenlecleucel — Tisagenlecleucel is single infusion.
  Other Names: CTL019

SUMMARY:
This is a multi-center, phase II study to determine the efficacy and safety of tisagenlecleucel in adult patients with relapsed or refractory FL.

DETAILED DESCRIPTION:
This single-arm, open label study had the following sequential phases: Screening, Pretreatment, Treatment and Follow-up. In the Pre-treatment phase, the patient could undergo bridging therapy (optional) and lymphodepleting (LD) chemotherapy. Treatment and Follow-up Phase included tisagenlecleucel infusion, and safety and efficacy follow-up for at least 24 months. For all the patients who received tisagenlecleucel infusion, additional survival follow-up was to be performed to determine survival status every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Refractory or relapsed Follicular Lymphoma (Grade 1, 2, 3A)
* Radiographically measurable disease at screening

Exclusion Criteria:

* Evidence of histologic transformation
* Follicular Lymphoma Grade 3B
* Prior anti-CD19 therapy
* Prior gene therapy
* Prior adoptive T cell therapy
* Prior allogeneic hematopoietic stem cell transplant
* Active CNS involvement by malignancy

Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2025-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (31):
- United States (9):
  - City of Hope National Medical Center, Duarte, California
  - UCSF Medical Center, San Francisco, California
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Uni of Chi Medi Ctr Hema and Onco, Chicago, Illinois
  - Univ of Kansas Hosp and Med Ctr, Kansas City, Kansas
  - Michigan Med University of Michigan, Ann Arbor, Michigan
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania Clinical, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Herston
- Novartis Investigative Site, Linz, Austria
- Novartis Investigative Site, Ghent, Belgium
- France (2):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
- Germany (3):
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Ulm
- Italy (2):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Milan, MI
- Japan (3):
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Sendai, Miyagi
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam, North Holland
  - Amsterdam UMC, locatie AMC, Amsterdam
- Novartis Investigative Site, Oslo, Norway
- Spain (2):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Madrid
- United Kingdom (2):
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Dreyling M, Fowler NH, Dickinson M, Martinez-Lopez J, Kolstad A, Butler J, Ghosh M, Popplewell L, Chavez JC, Bachy E, Kato K, Harigae H, Kersten MJ, Andreadis C, Riedell PA, Ho PJ, Perez-Simon JA, Chen AI, Nastoupil LJ, von Tresckow B, Maria Ferreri AJ, Teshima T, Patten PEM, McGuirk JP, Petzer AL, Offner F, Viardot A, Zinzani PL, Malladi R, Paule I, Zia A, Awasthi R, Han X, Germano D, O'Donovan D, Ramos R, Maier HJ, Masood A, Thieblemont C, Schuster SJ. Durable response after tisagenlecleucel in adults with relapsed/refractory follicular lymphoma: ELARA trial update. Blood. 2024 Apr 25;143(17):1713-1725. doi: 10.1182/blood.2023021567. PMID 38194692
- [Derived] Salles G, Schuster SJ, Dreyling M, Fischer L, Kuruvilla J, Patten PEM, von Tresckow B, Smith SM, Jimenez-Ubieto A, Davis KL, Anjos C, Chu J, Zhang J, Lobetti Bodoni C, Thieblemont C, Fowler NH, Dickinson M, Martinez-Lopez J, Wang Y, Link BK. Efficacy comparison of tisagenlecleucel vs usual care in patients with relapsed or refractory follicular lymphoma. Blood Adv. 2022 Nov 22;6(22):5835-5843. doi: 10.1182/bloodadvances.2022008150. PMID 35973192
- [Derived] Fowler NH, Dickinson M, Dreyling M, Martinez-Lopez J, Kolstad A, Butler J, Ghosh M, Popplewell L, Chavez JC, Bachy E, Kato K, Harigae H, Kersten MJ, Andreadis C, Riedell PA, Ho PJ, Perez-Simon JA, Chen AI, Nastoupil LJ, von Tresckow B, Ferreri AJM, Teshima T, Patten PEM, McGuirk JP, Petzer AL, Offner F, Viardot A, Zinzani PL, Malladi R, Zia A, Awasthi R, Masood A, Anak O, Schuster SJ, Thieblemont C. Tisagenlecleucel in adult relapsed or refractory follicular lymphoma: the phase 2 ELARA trial. Nat Med. 2022 Feb;28(2):325-332. doi: 10.1038/s41591-021-01622-0. Epub 2021 Dec 17. PMID 34921238

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 90 patients were planned, 98 patients were enrolled and 97 patients were infused with tisagenlecleucel.
Pre-assignment Details: During the Screening phase and prior to enrolment into the study, a patient's white blood cells were collected via leukapheresis.
Period: Overall Study
Arm/Group | CTL019
Started (Started = enrolled and entered pre-treatment phase) | 98
Treated (Treated = infused with tisagenlecleucel) | 97
Discontinued Prior to Infusion With Tisagenlecleucel | 1
Completed (Completed = Ongoing/in follow-up) | 80
Not Completed | 18
Not completed — Death | 7
Not completed — Physician Decision | 5
Not completed — Subject decision | 5
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Enrolled Set: All the patients who were enrolled in this study. Enrollment is defined as the point at which the patient meets all inclusion/exclusion criteria, and the patients' leukapheresis product was received and accepted by the manufacturing facility.
Arm/Group | CTL019
Number analyzed (Participants) | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (10.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 74
  Asian: Japanese | 9
  Asian: Indian | 2
  Asian: Missing (participants identified as Asian but with no other details provided) | 2
  Black or African American | 1
  Missing (No race/ethnicity provided) | 10

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate (CRR) Per Independent Review Committee (IRC) Assessment
Description: Complete response rate was defined as the percentage of participants with a best overall response (BOR) of complete response (CR) recorded from tisagenlecleucel infusion until progressive disease or start of new anticancer therapy, whichever came first. CRR was determined by an independent review committee (IRC) and was based on Lugano 2014 classification response criteria. The radiological response is first obtained from CT and PET studies according to the Lugano 2014 criteria. CT response is based on anatomical measurements of index/non-index/new lesions and spleen length. The possible response outcomes are complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD). PET response based on a 5-point scale (5PS) or Deauville score. The possible outcomes for PET response are complete metabolic response (CMR), partial metabolic response (PMR), no metabolic response (NMR), or progressive metabolic disease (PMD).
Time Frame: 1 year
Population: Efficacy analysis set (EAS): All the patients who received tisagenlecleucel, and had measurable disease at baseline per IRC. Non-measurable disease at baseline is defined as absence of index lesion at baseline disease evaluation (i.e. no disease at baseline).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CTL019
Number analyzed (Participants) | 94
Percentage of participants | 69.1 [58.8 to 78.3]

2. Secondary Outcome: Overall Response Rate (ORR) Per IRC Assessment
Description: Overall response rate is defined as the percentage of participants with a best overall disease response of complete response (CR) or partial response (PR). Response was evaluated per Lugano 2014 classification response criteria. The radiological response is first obtained from CT and PET studies according to the Lugano 2014 criteria. CT response is based on anatomical measurements of index/non-index/new lesions and spleen length. The possible response outcomes are complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD). PET response based on a 5-point scale (5PS) or Deauville score. The possible outcomes for PET response are complete metabolic response (CMR), partial metabolic response (PMR), no metabolic response (NMR), or progressive metabolic disease (PMD).
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage or participants
Arm/Group | CTL019
Number analyzed (Participants) | 94
Percentage or participants | 86.2 [77.5 to 92.4]

3. Secondary Outcome: Duration of Response (DOR) Per IRC
Description: Duration of response (DOR) applied only to participants whose best overall disease response was CR or PR. It is defined as the time from the date of first documented disease response (CR or PR) to the date of first documented progression or death due to follicular lymphoma (FL).
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2026-05

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Time from tisagenlecleucel infusion to first documented disease progression or death due to any cause
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2026-05

5. Secondary Outcome: Overall Survival (OS)
Description: Time from tisagenlecleucel infusion to death due to any cause
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2026-05

6. Secondary Outcome: Tisagenlecleucel Transgene Concentration
Description: Transgene concentration as detected by qPCR in target tissue
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2026-05

7. Secondary Outcome: Cmax; Cellular Kinetic Parameter of Tisagenlecleucel
Description: The maximum (peak) observed in peripheral blood or other body fluid drug concentration after single dose administration (% or copies/ µg)
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2026-05

8. Secondary Outcome: Tmax; Cellular Kinetic Parameter of Tisagenlecleucel
Description: The time to reach maximum (peak) peripheral blood or other body fluid drug concentration after single dose administration (days)
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2026-05

9. Secondary Outcome: AUC0-28; Cellular Kinetic Parameter of Tisagenlecleucel
Description: The AUC from time zero to day 28, in peripheral blood (%*days or days*copies/ µg)
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2026-05

10. Secondary Outcome: AUC0-84d; Cellular Kinetic Parameter of Tisagenlecleucel
Description: The AUC from time zero to day 84, in peripheral blood (%*days or days*copies/ µg)
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2026-05

11. Secondary Outcome: T1/2; Cellular Kinetic Parameter of Tisagenlecleucel
Description: The half-life associated with the elimination phase slope of a semi logarithmic concentration-time curve (days) in peripheral blood
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2026-05

12. Secondary Outcome: Tlast; Cellular Kinetic Parameter of Tisagenlecleucel
Description: The last observed measureable timepoint after dose administration
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2026-05

13. Secondary Outcome: Summary of Exposure of CD3+ Tisagenlecleucel Cells in Peripheral Blood
Description: In vivo cellular kinetics of CD3+ tisagenlecleucel cells detected by flow cytometry
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2026-05

14. Secondary Outcome: Humoral Immunogenicity
Description: Antibody titers specific to the tisagenlecleucel molecule prior to and following infusion.
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2026-05

15. Secondary Outcome: Cellular Immunogenicity
Description: Presence of T lymphocytes activated by the tisagenlecleucel protein
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2026-05

16. Secondary Outcome: Summary Scores of PRO Measured by SF-36v2 Quality of Life Questionnaire
Description: Effect of tisagenlecleucel therapy on Patient reported outcomes
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2026-05

17. Secondary Outcome: Summary Scores of PRO Measured by EQ-5D-3L Quality of Life Questionnaire
Description: Effect of tisagenlecleucel therapy on Patient reported outcomes
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2026-05

18. Secondary Outcome: Summary Scores of PRO Measured by FACT-Lym Quality of Life Questionnaire
Description: Effect of tisagenlecleucel therapy on Patient reported outcomes
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2026-05

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the post-infusion period (starting at the day of infusion until the end of the study), up to maximum duration of 24 months for each patient.
Description: AE Description: Any sign or symptom that occurs during the post-infusion period (starting at the day of first infusion of CTL019 until the end of the study).
Arm/Group | CTL019
All-Cause Mortality (participants affected / at risk) | 7/97
Serious Adverse Events (participants affected / at risk) | 42/97
Other Adverse Events (participants affected / at risk) | 94/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CTL019 (N=97)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 2
Ventricular fibrillation (Cardiac disorders) | 1
Blindness (Eye disorders) | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 1
Glossitis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Catheter site haemorrhage (General disorders) | 1
Pyrexia (General disorders) | 3
Cytokine release syndrome (Immune system disorders) | 19
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1
Bacteraemia (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
COVID-19 pneumonia (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Human herpesvirus 6 encephalitis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Parainfluenzae virus infection (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 8
Pneumonia haemophilus (Infections and infestations) | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1
Pseudomonal bacteraemia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2
Platelet count decreased (Investigations) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Encephalopathy (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CTL019 (N=97)
Anaemia (Blood and lymphatic system disorders) | 24
Febrile neutropenia (Blood and lymphatic system disorders) | 8
Leukopenia (Blood and lymphatic system disorders) | 8
Lymphopenia (Blood and lymphatic system disorders) | 8
Neutropenia (Blood and lymphatic system disorders) | 41
Thrombocytopenia (Blood and lymphatic system disorders) | 19
Abdominal pain (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 21
Nausea (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 8
Asthenia (General disorders) | 6
Chills (General disorders) | 7
Fatigue (General disorders) | 16
Pyrexia (General disorders) | 16
Cytokine release syndrome (Immune system disorders) | 30
Hypogammaglobulinaemia (Immune system disorders) | 14
Nasopharyngitis (Infections and infestations) | 6
Sinusitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 7
Lymphocyte count decreased (Investigations) | 9
Neutrophil count decreased (Investigations) | 17
Platelet count decreased (Investigations) | 10
SARS-CoV-2 test negative (Investigations) | 6
Weight decreased (Investigations) | 6
White blood cell count decreased (Investigations) | 21
Decreased appetite (Metabolism and nutrition disorders) | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 8
Hypophosphataemia (Metabolism and nutrition disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Back pain (Musculoskeletal and connective tissue disorders) | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 7
Headache (Nervous system disorders) | 24
Insomnia (Psychiatric disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 6
Hypertension (Vascular disorders) | 5
Hypotension (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e. data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT03568461/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT03568461/SAP_001.pdf